CLINICAL TRIAL: NCT06666829
Title: Innovative Paths to Paediatric Care: A Multicenter Study on the Efficacy of Multi-Domain Technological and Robotic Rehabilitation.
Brief Title: Multicenter Study That Offers New Solutions for Paediatric Rehabilitation by Proposing a Rehabilitation Plan Based on Each Child's Needs Using New Technological and Robotic Devices, Combined Among Them.
Acronym: MultiTECHChild
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: IRCCS Eugenio Medea (Other); Fondazione Don Carlo Gnocchi Onlus (Other); Fondazione Mondino (Other); Istituto Giannina Gaslini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNC0000007; PNC0000007 - Fit4MedRob (Other: Ministry of University and Research of Italy)
Record Dates: First submitted 2024-10-23; First posted 2024-10-31 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-10

CONDITIONS: Neuromotor Impairments
Keywords: Children; Multidomain; Robotic rehabilitation; Technological rehabilitation; Innovative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multidomain treatment group (Experimental): Participant will undergo a Multidomain rehabilitation treatment using the combination of two or more innovative technological and robotic devices.This will also be associated with the conventional rehabilitation
  Interventions: Other: Multidomain intervention
- Single domain treatment group (Active Comparator): Participant will undergo a Single domain rehabilitation treatment using only one innovative technological or robotic device.This will also be associated with the conventional rehabilitation
  Interventions: Device: Single domain intervention

INTERVENTIONS:
Other: Multidomain intervention — treatment plan using combination of more than one technological or robotic devices, choosing from: Virtual Reality Rehabilitation System (VRSS), Khymeia TR; HomeKIT Khymeia; VRSS Khymeia EVO; Myro® Tyromotion; Diego Tyromotion; Tyrostation Tyromotion; Pablo® Tyromotion; Amadeo Tyromotion; Lexo® Tyromotion; Humaware MObile RoboT for upper Limb NeurOortho Rehabilitation (MOTORE); Humanware Upper Limb TRAcker(ULTRA+); Gloreha Sinfonia plus; C-Mill Motek; Gait Real Time Analysis Laboratory (GRAIL) Motek Medical; Nirvana BTS; Agilik; Armeo Spring pediatrico Hocoma; Lokomat ® Hocoma; Hand Tutor, Leg Tutor, Arm Tutor (MediTouch); Care Lab; Dessintey IVS3; Rehacom Hasomed; Hunova; GEO System (Kineo).
  In this way, the child will be taken care of holistically, considering their needs from a motor, cognitive, and speech therapy perspective. The treatment plan will also include a conventional multi-level rehabilitation program.
  Arms: Multidomain treatment group
Device: Single domain intervention — Treatment plan using only one of these technological or robotic device:
  Virtual Reality Rehabilitation System (VRSS), Khymeia TR; HomeKIT Khymeia; VRSS Khymeia EVO; Myro® Tyromotion; Diego Tyromotion; Tyrostation Tyromotion; Pablo® Tyromotion; Amadeo Tyromotion; Lexo® Tyromotion; Humaware MObile RoboT for upper Limb NeurOortho Rehabilitation (MOTORE); Humanware Upper Limb TRAcker(ULTRA+); Gloreha Sinfonia plus; C-Mill Motek; Gait Real Time Analysis Laboratory (GRAIL) Motek Medical; Nirvana BTS; Agilik; Armeo Spring pediatrico Hocoma; Lokomat ® Hocoma; Hand Tutor, Leg Tutor, Arm Tutor (MediTouch); Care Lab; Dessintey IVS3; Rehacom Hasomed; Hunova; GEO System (Kineo).
  Technological rehabilitation will focus on the main specific need for the child, it'll be chosen individually. The treatment plan will also include a conventional multi-level rehabilitation program.
  Arms: Single domain treatment group

SUMMARY:
The goal of this clinical trial is to demonstrate the efficacy of multi domain robotic and technological rehabilitation on everyday life and satisfaction in children with neuromotor conditions. The main questions it aims to answer are:

* Will we have significant changes using the COPM in children taking part in the sperimental group?
* The children who will undergo the multidomain treatment will also experience functional improvements in individual areas?
* Thy type of treatment will improve motivation, active participation and satisfaction in children?

Researcher will compare the multidomain treatment to standard care proposed by the included clinical centers: single domain rehabilitation with one innovative device. Both groups will undergo also conventional multidomain therapy.

This will be done to see if using a holistic approach, and including every need of the child in the rehabilitation plan, can lead to greater improvements in quality of life compared to the control group.

Participant will:

* Be evaluated 3 times with clinical outcome measures
* Take part in a rehabilitation program, at least 20 x 2hours sessions treatment, organized in:

  * 4 weeks, 5 times per week
  * 7 weeks, 3 times per week

DETAILED DESCRIPTION:
* The sample size was determined considering the primary outcome (the change in COPM): the superiority of robotic treatment compared to conventional treatment; a power of 80%; a number of groups equal to 2; a number of measurements equal to 3; and an effect size of 0.1. Based on these parameters, a sample size of 162 patients (81 per group) is obtained. Additionally, considering a dropout rate of 20%, a total sample size of 194 patients is required.
* For each recruited subject, a specific checklist (CRF) will be completed to collect the demographic, clinical, and technological data required by the study. All collected data will be pseudonymized (using a technique that modifies and masks personal and sensitive data to prevent it from being directly and easily attributed to an individual), in accordance with current privacy regulations. This will allow for regular monitoring of the study's progress, particularly regarding the number of subjects enrolled and recruited in the different phases, the evaluation tests conducted, adherence to the study, and the treatment protocols implemented.
* A high adherence to the study is anticipated, especially if the children involved receive treatment during the care period in rehabilitation facilities, in compliance with current regulations. To ensure the quality and consistency of the intervention, a careful assessment of adherence will be conducted. This assessment will be carried out by an independent team of clinical reviewers, who will regularly monitor treatment sessions. The reviewers will then implement targeted strategies to maintain and improve adherence, including periodic training sessions for the staff involved and timely feedback directed to the therapists in both study groups. A diary will also be maintained regarding the treatments performed by each patient to monitor adherence to the proposed treatment.
* Regarding the collection of data obtained from standardized clinical evaluations, each subject will be assigned a numeric ID code in accordance with current privacy regulations, allowing for the preservation and sharing of data in a completely anonymous form with other participating centers. The list linking the assigned code to each child's name will be kept by the principal investigator and stored in a locked cabinet. Only the principal investigator and other researchers involved in the project will have access to this information.

Similarly, information obtained during the rehabilitation phase from technological tools will be stored and shared with other participating centers in a completely anonymous manner, using the same numeric code previously defined. The data collected throughout the study, excluding the subject's name, will be recorded, processed, and stored for at least seven (7) years after the conclusion of the study, along with the assigned code, on password-protected hard drives stored in a physically secured location or within protected electronic archives (Research Electronic Data Capture (RedCap)), accessible only to the principal investigator and authorized researchers. After seven years, the data will be destroyed.

All collected information will not be processed or used for purposes other than those indicated in the study's objectives, nor for direct profit, and will not be communicated or transferred to unauthorized third parties.

Personal data will be collected and processed in accordance with the principle of data minimization and in compliance with all general principles outlined in Article 5 of the GDPR. Data, particularly personal and health-related data, will be processed only to the extent necessary in relation to the objectives of the trial, in accordance with EU Regulation 2016/679 (GDPR) and Legislative Decree No. 101 of August 10, 2018.

At the time of data collection, whether obtained from standardized clinical evaluations or from device reports, the Data Controllers will ensure that the collected data is pseudonymized by identifying the recruited subjects with codes or adopting other solutions compliant with point 5.4 of the Privacy Authority Provision No. 146/2019. The use of encryption techniques allows for the storage and processing of the data subject's information in a way that prevents identification by any external person. Only the Project Manager at each center and authorized personnel can link each code to the name of the participating subject.

•Regarding any events to be reported, the mode and timing of reporting will adhere to the obligations imposed by EU Regulation 2017/745 (Article 80) and the MDCG Guideline 2020-10/1 ("Safety reporting in clinical investigations of medical devices under Regulation (EU) 2017/745").

A specific insurance policy will be established, which will be activated immediately before the start of the clinical trial. Insurance quotes have been requested and are currently under evaluation. The policy will comply with the provisions of the Ministerial Decree of July 14, 2009, which guarantees specific coverage for damages caused to subjects by the trial activities throughout its duration, covering the civil liability of the investigator and the sponsor, without excluding damages unintentionally caused as a result of an accidental event and/or attributable to negligence, imprudence, or incompetence.

•The collected data will be presented using descriptive statistics, such as mean and standard deviation for numerical variables, and percentages for categorical variables.

The population will be defined to include patients in the multidomain treatment group or the control group (monodomain). The analyzable population will be defined by excluding patients who are not eligible for entry and those who do not receive the full treatment (due to treatment interruption for any reason). The primary endpoint at the end of treatment will be compared between the two treatment groups.

For the primary outcome, a planned subgroup analysis will be conducted to assess the presence of treatment effect modifiers. Continuous secondary outcomes will be analyzed in the population. All tests will be two-tailed with a significance level of 5%, and effect estimates will include a 95% confidence interval (CI).

Categorical outcomes will be reported as proportions with 95% CIs and compared using appropriate statistical tests. Similar analysis will be conducted to demonstrate any improvement in parameters measured during the follow-up (T2). This analysis will include subjects who completed the treatment, representing the population to be studied in the months following the completion of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of developmental disorder and/or disability, either congenital or acquired;
* Age between 5 and 21 years at the time of recruitment;
* Verbal and/or non-verbal reasoning abilities > 70 or > 5th percentile, as assessed by standardized tests such as Colored Progressive Matrices (CPM), WISC-IV or WISC-V, WPPSI-III or WPPSI-IV, Leiter-3, Griffiths III.

Exclusion Criteria:

* Presence of severe comorbidities and/or behavioral/cognitive disorders that prevent adequate patient compliance with both conventional and robotic rehabilitation treatment (severe intellectual disability);
* Uncontrolled epilepsy;
* Presence of severe sensory deficits;
* Patients who have undergone orthopedic functional surgery or rhizotomy and/or botulinum toxin treatment in the last 6 months;
* Involvement of the peripheral nervous system

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 194 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  Assessment tool used in occupational therapy to evaluate an individual's performance and satisfaction in both daily and personal activities. The COPM focuses on activities that are meaningful to the assessed person, allowing them to identify areas where they wish to improve their abilities or participation. This tool helps therapists better understand their patients' needs and desires, enabling them to plan targeted therapeutic interventions to enhance their quality of life and overall well-being.

SECONDARY OUTCOMES:
Melbourne Assessment-2 (MA2) | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  A standardized, valid, and reliable tool for assessing the quality of upper limb movement in children with neurological deficits aged between 2.5 and 15 years. The MA2 measures four elements of movement quality: range of motion, accuracy, dexterity, and fluidity. It consists of 14 items for reaching, grasping, releasing, and manipulating simple objects. For each item the examiner gives a score ranging from 0 to 4, higher score corresponds to better performance.A raw score and percentage score are provided for each of the four sections, which will be analyzed separately. The test is administered by video recording the child's performance, which will be evaluated later by the examiner.
ABILHAND-Kids. | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  The ABILHAND-Kids is a brief questionnaire that measures 21 key bimanual daily activities. The score is assigned by a parent based on the difficulty the child has in performing the requested activity on a daily basis, using a 3-point scale (impossible, difficult, easy). The response scores are entered into a Rasch model to obtain a continuous score representing the child's level of manual ability. A higher score indicates greater manual skill and autonomy.
  It has been validated in children with Cerebral Palsy aged 6 to 15 years, showing good validity (R=0.94) and good reproducibility over time (R=0.91).
Gross Motor Function Measure-88 (GMFM-88). | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  The GMFM-88 is an assessment tool used to measure gross motor ability in children with motor disabilities, particularly those affected by cerebral palsy. It is designed to evaluate motor function in areas such as positioning, movement, trunk control, and locomotion. The GMFM-88 consists of a series of 88 items divided into five dimensions (A, B, C, D, E), with each item rated on a 4-point scale (0-3) that reflects the child's level of ability for that specific task. Single scores are summed to obtain a partial score for each dimension. The partial scores are then combined to calculate a total score, represented as a percentage that reflects the child's overall performance in gross motor skills. A higher score indicates better gross motor function.
Six Minutes Walking Test (6MWT) | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  A test used to assess walking endurance in children with cerebral palsy. During the test, the child is encouraged to walk as much as possible for a period of six minutes along a standardized pathway. The score is assigned based on the total distance covered in six minutes and the distance covered separately in each minute, expressed in meters. This distance is then interpreted according to normative tables that vary by age, gender, and sometimes health status to determine if the result is adequate, below average, or above average. This test provides valuable information about the child's level of endurance during walking and can be used to monitor progress over time and evaluate the effectiveness of therapeutic interventions.
NEPSY-II inibition and auditory attention subtest | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  INIBITION: It assesses the ability to inhibit automatic responses in favor of new ones and to switch from one type of response to another. It is divided into three conditions: naming, inhibition, and switching. For each condition, both accuracy and speed are obtained, with standardized scores ranging from 1 to 19. Higher scores indicate better performance.
  AUDITORY ATTENTION: It assesses the ability to analyze and select target stimuli among distractors using auditory material. The score is indicated in percentiles.
Leiter 3- Sustained attention subtest | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  It evaluates sustained visual attention and consists of repetitive barrage tasks to be completed within a predefined time. The number of correctly selected target items is recorded. Raw scores range from 0 to 217, while standardized scores range from 1 to 19. Higher scores indicate better performance.
VMI | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  It is a pencil-and-paper test used to determine the level of integration between visual and motor systems. The child is asked to copy various geometric shapes presented on the paper within a certain timeframe. The number of correctly reproduced figures is recorded and then converted into standardized scores. Raw scores range from 0 to 27, with higher scores indicating better performance.
Tower of London (ToL) | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  It is a test useful for studying and measuring planning skills. The child must place three marbles (red, green, and blue) on a stand consisting of three pegs of different lengths in various configurations, following specific rules.
  The total score is a combination of the number of problems solved correctly, the number of moves used, the errors made, and the time taken (if included). A higher score indicates greater planning and problem-solving abilities.
BVL 4-12 | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  The BVL 4-12 battery systematically evaluates phonological, lexical, semantic, pragmatic, and discourse skills through tasks of oral production, comprehension, and repetition in children aged 4 to 12 years, highlighting any communication and language disorders.
  It's composed of 18 tasks each of which contains a different number of items; for each item a score from 0 to 1 is given. Scores are summed up to have a final score for each area, raw scores are transformed into z standardized scores according to normative data.
  Higher score correspond to better performance.
BVN 12-18 language, reading and writing subtest | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  The BVN 12-18 battery evaluates language reading, writing, and in adolescents aged 12 to 18 years.
  This part is composed of 7 tasks each of which contains a different number of items; for each item a score from 0 to 1 is given. Except for reading items where reading speed and accuracy are evaluated in syllables/seconds and error rate.
  Scores are summed up to have a final score for each area, raw scores are transformed into z standardized scores according to normative data.
  Higher score correspond to better performance.
MT-3 tests | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  Tests aimed at evaluating reading skills and text comprehension for primary and lower secondary school classes.
  Reading speed and accuracy were evaluated by presenting children with a text and asking them to read it. Reading speed was measured in syllables per second (s/s). The error rate was calculated using the total number of words read.
  For text comprehension we ask the child to read 2 texts and answer questions, for each of it a score from 0 to 1 is given and then summed; higher score corresponds to better performance.
  Raw scores are transformed into z standardized scores according to normative data.
BVSCO-3 | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  BVSCO-3 tests measures the child's orthographic skills in terms of percentages of spelling errors made in dictation text task. Raw scores are transformed into z standardized scores according to normative data
HTA Questionnaires | Up to 7 weeks after the baseline (T1)
  Questionnaires to be administered to various stakeholders (child, caregivers, and therapist) aimed at assessing the usability and acceptability of the proposed treatment. They will be constructed ad hoc based on specific aspects.
3D Gait Analysis: Joint kinematics | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  Joint angles: measured throughout the gait cycle at the hip, knee, and ankle. Range of Motion (ROM): assessed for the lower limbs and trunk to evaluate the amplitude of joint movements.
  Joint angles are measured in degrees.
3D Gait Analysis: Kinetics - Ground Reaction Force | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  Ground Reaction Force (GRF): assessed in vertical, anteroposterior, and mediolateral directions to understand the forces exerted by the ground on the body.
3D Gait Analysis: Kinetics - Joint moments | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  Joint moments: calculated at the hip, knee, and ankle to evaluate the forces acting on these joints throughout the gait cycle, expressed in Newton-meters, normalized by body weight in kilograms.
3D Gait Analysis: Kinetics - Joint power | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  Joint power: power generated and absorbed at the joints during gait, expressed in watts, normalized by body weight in kilograms
3D Gait Analysis: Spatiotemporal parameters | baseline(T0), up to 7 weeks (T1) and 2 months after the end of the training (T2)
  Step and stride length: the distance covered per step and per full gait cycle, measured in meters.
  Duration of step and stride: time taken for each step and each complete stride, measured in seconds and as percentages of the gait cycle.
  Cadence: number of steps per minute. Walking speed: velocity of walking, which is a key indicator of gait efficiency.
  Stance and swing phase durations: the time spent in stance (foot in contact with the ground) and swing phases during the gait cycle.

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - IRCCS Giannina Gaslini, Genova, Genova
  - IRCCS Eugenio Medea, Bosisio Parini, Lecco
  - Fondazione Don Gnocchi IRCCS centro "Santa Maria Nascente", Milan, Milano
  - IRCCS Istituto Neurologico Naz.le C.Mondino, Pavia, Pavia
  - IRCCS Fondazione Stella Maris, Calambrone, Pisa
  - Fondazione Don Gnocchi IRCCS centro "S.Maria al Mare", Salerno, Salerno

IPD SHARING:
Plan to Share IPD: No